CLINICAL TRIAL: NCT00679809
Title: Safety, Fatigue, and Continuity in the ICU: a Pragmatic Mixed-methods Study
Brief Title: Safety, Fatigue, and Continuity in the Intensive Care Unit (ICU)
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Christopher Parshuram, Staff Physician, The Hospital for Sick Children
Other Study IDs: 1000011945
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Fatigue
Keywords: Resident; Safety; Fatigue; Continuity; ICU
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to describe the features of continuity and quantify fatigue in three ICU resident work schedules, estimate the frequency of preventable adverse events, and inform the design and demonstrate the feasibility of a future multi-centre study.

DETAILED DESCRIPTION:
The overall goal of our research is to describe the optimal scheduling pattern for frontline physicians working in ICUs. Our hypothesis is that call schedule associated reductions in fatigue are counterbalanced by reductions in continuity, resulting in no change in the safety of patients.

This is a prospective before-after, two-centre study using a mixed-methods design. We will apply 3 work schedules, each for a period of 2 months over a 6 month period in the adult medical-surgical ICUs at two university affiliated hospitals in Toronto. In this mixed methods approach, quantitative and qualitative data will be collected concurrently, analysed separately, and their results compared, to produce an integrated interpretation of the impact of work schedule on the relationship between continuity and fatigue.

This will evaluate healthcare continuity and fatigue, describe adverse events in ICUs, identify the two best resident schedules for subsequent comparison, and demonstrate the feasibility of a future multi-centre study of physician scheduling.

ELIGIBILITY:
Inclusion Criteria:

* All residents at participating ICUs starting a rotation in Fall 2008
* Staff members supervising and/or working with participating residents
* Patients/family members under the care of the participating residents
* Patients admitted to participating ICUs

Exclusion Criteria:

* Lack of informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Residents will be on their 2-month ICU rotations at one of two university affiliated hospitals in Toronto medical-surgical ICU. Residents in these ICU rotations are from internal medicine, surgery, emergency medicine and anesthesia training programs, and are supported by 2-3 critical care fellows, and 1 staff physician
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2008-10; Primary Completion 2009-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Fatigue | 6 months
Continuity of patient care | 6 months

SECONDARY OUTCOMES:
Adverse events | 6 months
Preventable adverse events | 6 months
Feasibility | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Chris Parshuram, MBChB, PhD, Principal Investigator — The Hospital for Sick Children; Jan Friedrich, MD, Principal Investigator — Unity Health Toronto; Thomas Stewart, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (3):
- Canada (3):
  - Mount Sinai Hospital, Toronto, Ontario
  - St Michael's Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

REFERENCES:
- [Derived] Parshuram CS, Amaral AC, Ferguson ND, Baker GR, Etchells EE, Flintoft V, Granton J, Lingard L, Kirpalani H, Mehta S, Moldofsky H, Scales DC, Stewart TE, Willan AR, Friedrich JO; Canadian Critical Care Trials Group. Patient safety, resident well-being and continuity of care with different resident duty schedules in the intensive care unit: a randomized trial. CMAJ. 2015 Mar 17;187(5):321-9. doi: 10.1503/cmaj.140752. Epub 2015 Feb 9. PMID 25667258